CLINICAL TRIAL: NCT00340353
Title: Procurement of Blood and Tissue From Patients With Primary and Metastatic Alveolar Soft Part Sarcoma and Blood From Healthy Controls for In Vitro and In Vivo Model Development
Brief Title: Collection of Alveolar Soft Part Sarcoma and Blood Specimens for Research
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999905138; 05-C-N138
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2012-04-12

CONDITIONS: Alveolar Soft Part Sarcoma; Sarcoma
Keywords: Gene Expression; Drug Sensitivity; TFE3; ASPL-TFE3; NOD-SCID Mice; Sarcoma; Alveolar Soft Part Sarcoma; ASPS
MeSH Terms: conditions — Sarcoma, Alveolar Soft Part; Sarcoma

SUMMARY:
Background:

Alveolar soft part sarcoma (ASPS) is a rare tumor.

ASPS is resistant to chemotherapy and radiation.

ASPS is characterized by slow growth.

Currently no in vitro or in vivo models of ASPS exist for use in experimental therapeutic studies or biological investigations.

Primary Objectives:

Acquisition of blood and tissue from patients with ASPS.

Acquisition of blood from healthy controls for comparison with blood from patients with ASPS. These control samples will be obtained from study NCI at Frederick Protocol OH99-C-N046.

Eligibility:

Subjects of any age with a diagnosis of primary or metastatic alveolar soft part sarcoma who are undergoing medically indicated surgery for their disease.

Design:

Patients with Alveolar Soft Part Sarcoma (ASPS) will be eligible for this study. Biopsy tissue will be obtained as an additional sample at the time of a medically indicated procedure. Blood sample may be collected at initial visit and follow-up visits. Specific risks will be described in a separate consent to be obtained at the time of the biopsy. Tumor samples and blood samples will be processed and/or stored for use in research efforts in the laboratory of Dr. David Vistica, National Cancer Institute, Frederick, MD. Additionally, blood samples will be obtained from healthy volunteers for comparison to patients with ASPS. These control samples will be obtained from the National Cancer Institute at Frederick Protocol OH99-C-N046.

DETAILED DESCRIPTION:
Background:

Alveolar soft part sarcoma (ASPS) is a rare tumor.

ASPS is resistant to chemotherapy and radiation.

ASPS is characterized by slow growth.

Currently no in vitro or in vivo models of ASPS exist for use in experimental therapeutic studies or biological investigations were generated under this protocol.

Additional models are needed to represent the heterogeneity of this disease.

Primary Objectives:

Acquisition of blood and tissue from patients with ASPS.

Acquisition of blood from healthy controls for comparison with blood from patients with ASPS. These control samples will be obtained from study NCI at Frederick Protocol OH99-C-N046.

Eligibility:

Subjects of any age with a diagnosis of primary or metastatic alveolar soft part sarcoma who are undergoing medically indicated surgery for their disease.

Design:

Patients with Alveolar Soft Part Sarcoma (ASPS) will be eligible for this study. Biopsy tissue will be obtained as an additional sample at the time of a medically indicated procedure. Blood sample may be collected at initial visit and follow-up visits. Specific risks will be described in a separate consent to be obtained at the time of the biopsy. Tumor samples and blood samples will be processed and/or stored for use in research efforts in the laboratory of Dr. Robert Shoemaker, National Cancer Institute, Frederick, MD. Additionally, blood samples will be obtained from healthy volunteers for comparison to patients with ASPS. These control samples will be obtained from the National Cancer Institute at Frederick Protocol OH99-C-N046.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects of any age with a diagnosis of primary or metastatic alveolar soft part sarcoma who are undergoing medically indicated surgery for their disease.

EXCLUSION CRITERIA:

None.

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 99999 (Estimated)
Dates: Start 2005-04-07; Study Completion 2012-04-12

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dean, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] CHRISTOPHERSON WM, FOOTE FW Jr, STEWART FW. Alveolar soft-part sarcomas; structurally characteristic tumors of uncertain histogenesis. Cancer. 1952 Jan;5(1):100-11. doi: 10.1002/1097-0142(195201)5:13.0.co;2-k. No abstract available. PMID 14886902